CLINICAL TRIAL: NCT01294995
Title: Phase 1 Study of Chinese Tea-flavor Liquor
Brief Title: Effect of Short-term Chinese Tea-flavor Liquor Consumption
Acronym: ESTCTFLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: Guizhou Meijiao Co., Ltd (Unknown)
Responsible Party: Department of Food Science and Nutrition, Department of Food Science and Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ST Chinese liquor study
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2010-10

CONDITIONS: Cardiovascular Diseases
Keywords: short term consumption; Chinese liquor; serum lipids; uric acid; inflammation biomarkers
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tea-flavor Liquor, taken with meal (Experimental): including 12 males and 11 females
  Interventions: Dietary Supplement: Tea-flavor Liquor
- Guizhou Meijiao Liquor, taken with meal (Placebo Comparator): including 11 males and 11 females
  Interventions: Dietary Supplement: Guizhou Meijiao Liquor

INTERVENTIONS:
Dietary Supplement: Tea-flavor Liquor — 30 mL of Tea-flavor Liquor(45% alcohol content)
  Arms: Tea-flavor Liquor, taken with meal
Dietary Supplement: Guizhou Meijiao Liquor — 30 mL of Guizhou Meijiao Liquor (45% alcohol content)
  Arms: Guizhou Meijiao Liquor, taken with meal

SUMMARY:
Human studies of Chinese liquor are sparse. The investigators hypothesize that short-term Chinese Tea-flavor liquor (TFL) consumption may be beneficial to inflammation biomarkers and CVD risk factors. Guizhou Meijiao Liquor (GML) is a traditional Chinese liquor, fermented from sorghum, corn, sticky rice, wheat and rice, while TFL is a novel Chinese liquor fermented from above 5 grains plus green tea.

Forty-five volunteers(23 males, 22 females) were selected to participate a paralleled randomized trial drinking 30 mL two kinds of Chinese liquors: TFL and GML respectively with meal every day for 28 days. Serums of volunteers were collected for analyzing serum lipids, inflammation biomarkers and CVD risk factors.

TFL could significantly decrease systolic blood pressure of males, but increase diastolic blood pressure of females. TFL could also decreased blood lipid of volunteers, especially for females. Both liquor significantly decrease serum uric acid and glucose in males and females. The effect of the two liquors on inflammation biomarkers were complicated and needs further research work.

TFL may possess more beneficial effect on CVD risk factors than GML probably because of the special fermentation products of green tea with other grains.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers

Exclusion Criteria:

* Subjects with a history of liver disease, diabetes, or heart disease
* Smokers

Ages: 23 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of food science and nutrition, Hangzhou, Zhejiang, China